CLINICAL TRIAL: NCT06433544
Title: Evaluating the Effects of Online Mindfulness Therapy on Pandemic Fatigue and Resilience Among Nurses in COVID-19 Quarantine Wards
Brief Title: Online Mindfulness Therapy for Pandemic Fatigue and Resilience in COVID-19 Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chimei Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11112-001
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Mindfulness; Nurses in COVID-19; Pandemic Fatigue; Resilience
Keywords: Online mindfulness; COVID-19 quarantine ward nurses; Pandemic fatigue; Resilience

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group will undergo a 6-week online mindfulness course (Experimental): The experimental group received a 6-week online mindfulness course, once a week for 90 minutes each session. Participants completed questionnaires before the course, at week 3, and at week 6.
  Interventions: Other: 6-week online mindfulness course
- Control group (No Intervention): General routine care

INTERVENTIONS:
Other: 6-week online mindfulness course — The experimental group received a 6-week online mindfulness course, once a week for 90 minutes each session.
  Arms: Experimental group will undergo a 6-week online mindfulness course

SUMMARY:
This study evaluates online mindfulness therapy's impact on pandemic fatigue and resilience in COVID-19 quarantine ward nurses. Sixty nurses were divided into experimental and control groups, with the experimental group receiving a 6-week online mindfulness course.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of online mindfulness therapy on reducing pandemic fatigue and enhancing resilience among nurses in COVID-19 quarantine wards. Using a repeated-measures quasi-experimental design, 60 nurses were divided into experimental and control groups. The experimental group participated in a 6-week online mindfulness course. Outcomes were measured using pandemic fatigue and resilience questionnaires at the pre-test , three weeks and after six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old.
* Nurses of COVID-19 dedicated wards and dedicated intensive care units.

Exclusion Criteria:

* Difficulty in attending
* less than 80% of the total number of online mindfulness therapy sessions

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Pandemic Fatigue | 6 weeks
  Use Lockdown/Pandemic Fatigue Scale (LFS) measure pandemic fatigue. The scale with a total of 10 items measures pandemic fatigue. The range of total scores of the scale is 10-50. It shows that pandemic fatigue increases as total points of the scale increase.

SECONDARY OUTCOMES:
Resilience | 6 weeks
  Use Connor-Davidson Resilience Scale (CD-RISC) measure individual resilience. The scale with a total of 25 items measures resilience. The range of total scores of the scale is 0-100. It shows that resilience increases as total points of the scale increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Chi Mei Medical Center, Tainan, 其他（非美國）, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afshari D, Nourollahi-Darabad M, Chinisaz N. Demographic predictors of resilience among nurses during the COVID-19 pandemic. Work. 2021;68(2):297-303. doi: 10.3233/WOR-203376. PMID 33492260
- [Background] Amutio A, Martinez-Taboada C, Delgado LC, Hermosilla D, Mozaz MJ. Acceptability and Effectiveness of a Long-Term Educational Intervention to Reduce Physicians' Stress-Related Conditions. J Contin Educ Health Prof. 2015 Fall;35(4):255-60. doi: 10.1097/CEH.0000000000000002. PMID 26953856
- [Background] Asuero AM, Queralto JM, Pujol-Ribera E, Berenguera A, Rodriguez-Blanco T, Epstein RM. Effectiveness of a mindfulness education program in primary health care professionals: a pragmatic controlled trial. J Contin Educ Health Prof. 2014 Winter;34(1):4-12. doi: 10.1002/chp.21211. PMID 24648359
- [Background] Barnett P, Barnett M, Borgueta E, Moreno JV, Watson J. COVID-19: An Organizational-theory-guided Holistic Self-caring and Resilience Project. J Holist Nurs. 2021 Dec;39(4):325-335. doi: 10.1177/08980101211007007. Epub 2021 Apr 16. PMID 33861185
- [Background] Barry KM, Woods M, Martin A, Stirling C, Warnecke E. A randomized controlled trial of the effects of mindfulness practice on doctoral candidate psychological status. J Am Coll Health. 2019 May-Jun;67(4):299-307. doi: 10.1080/07448481.2018.1515760. Epub 2018 Nov 2. PMID 30388950
- [Background] Baskin RG, Bartlett R. Healthcare worker resilience during the COVID-19 pandemic: An integrative review. J Nurs Manag. 2021 Nov;29(8):2329-2342. doi: 10.1111/jonm.13395. Epub 2021 Jul 9. PMID 34182609
- [Background] Bazarko D, Cate RA, Azocar F, Kreitzer MJ. The Impact of an Innovative Mindfulness-Based Stress Reduction Program on the Health and Well-Being of Nurses Employed in a Corporate Setting. J Workplace Behav Health. 2013 Apr;28(2):107-133. doi: 10.1080/15555240.2013.779518. PMID 23667348
- [Background] Buleon C, Minehart RD, Fischer MO. Protecting healthcare providers from COVID-19 through a large simulation training programme. Br J Anaesth. 2020 Nov;125(5):e418-e420. doi: 10.1016/j.bja.2020.07.044. Epub 2020 Aug 5. No abstract available. PMID 32828493
- [Background] Cai Z, Cui Q, Liu Z, Li J, Gong X, Liu J, Wan Z, Yuan X, Li X, Chen C, Wang G. Nurses endured high risks of psychological problems under the epidemic of COVID-19 in a longitudinal study in Wuhan China. J Psychiatr Res. 2020 Dec;131:132-137. doi: 10.1016/j.jpsychires.2020.09.007. Epub 2020 Sep 14. PMID 32971356
- [Background] Catania G, Zanini M, Hayter M, Timmins F, Dasso N, Ottonello G, Aleo G, Sasso L, Bagnasco A. Lessons from Italian front-line nurses' experiences during the COVID-19 pandemic: A qualitative descriptive study. J Nurs Manag. 2021 Apr;29(3):404-411. doi: 10.1111/jonm.13194. Epub 2020 Nov 15. PMID 33107657
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Creswell JD, Lindsay EK, Villalba DK, Chin B. Mindfulness Training and Physical Health: Mechanisms and Outcomes. Psychosom Med. 2019 Apr;81(3):224-232. doi: 10.1097/PSY.0000000000000675. PMID 30806634
- [Background] Croghan IT, Chesak SS, Adusumalli J, Fischer KM, Beck EW, Patel SR, Ghosh K, Schroeder DR, Bhagra A. Stress, Resilience, and Coping of Healthcare Workers during the COVID-19 Pandemic. J Prim Care Community Health. 2021 Jan-Dec;12:21501327211008448. doi: 10.1177/21501327211008448. PMID 33834900
- [Background] Cuadrado E, Maldonado MA, Tabernero C, Arenas A, Castillo-Mayen R, Luque B. Construction and Validation of a Brief Pandemic Fatigue Scale in the Context of the Coronavirus-19 Public Health Crisis. Int J Public Health. 2021 Aug 30;66:1604260. doi: 10.3389/ijph.2021.1604260. eCollection 2021. PMID 34566554
- [Background] de Vibe M, Solhaug I, Tyssen R, Friborg O, Rosenvinge JH, Sorlie T, Bjorndal A. Mindfulness training for stress management: a randomised controlled study of medical and psychology students. BMC Med Educ. 2013 Aug 13;13:107. doi: 10.1186/1472-6920-13-107. PMID 23941053
- [Background] Dharra S, Kumar R. Promoting Mental Health of Nurses During the Coronavirus Pandemic: Will the Rapid Deployment of Nurses' Training Programs During COVID-19 Improve Self-Efficacy and Reduce Anxiety? Cureus. 2021 May 24;13(5):e15213. doi: 10.7759/cureus.15213. PMID 34178532
- [Background] Dincer B, Inangil D. The effect of Emotional Freedom Techniques on nurses' stress, anxiety, and burnout levels during the COVID-19 pandemic: A randomized controlled trial. Explore (NY). 2021 Mar-Apr;17(2):109-114. doi: 10.1016/j.explore.2020.11.012. Epub 2020 Dec 3. PMID 33293201
- [Background] Duarte J, Pinto-Gouveia J. Effectiveness of a mindfulness-based intervention on oncology nurses' burnout and compassion fatigue symptoms: A non-randomized study. Int J Nurs Stud. 2016 Dec;64:98-107. doi: 10.1016/j.ijnurstu.2016.10.002. Epub 2016 Oct 8. PMID 27744228
- [Background] Ducar DM, Penberthy JK, Schorling JB, Leavell VA, Calland JF. Mindfulness for healthcare providers fosters professional quality of life and mindful attention among emergency medical technicians. Explore (NY). 2020 Jan-Feb;16(1):61-68. doi: 10.1016/j.explore.2019.07.015. Epub 2019 Aug 6. PMID 31471216
- [Background] Duchemin AM, Steinberg BA, Marks DR, Vanover K, Klatt M. A small randomized pilot study of a workplace mindfulness-based intervention for surgical intensive care unit personnel: effects on salivary alpha-amylase levels. J Occup Environ Med. 2015 Apr;57(4):393-9. doi: 10.1097/JOM.0000000000000371. PMID 25629803
- [Background] Elliott M, Khallouf C, Hirsch J, de Camps Meschino D, Zamir O, Ravitz P. Novel Web-Based Drop-In Mindfulness Sessions (Pause-4-Providers) to Enhance Well-Being Among Health Care Workers During the COVID-19 Pandemic: Descriptive and Qualitative Study. JMIR Form Res. 2024 Mar 14;8:e43875. doi: 10.2196/43875. PMID 38180869
- [Background] Fernandez-Castillo RJ, Gonzalez-Caro MD, Fernandez-Garcia E, Porcel-Galvez AM, Garnacho-Montero J. Intensive care nurses' experiences during the COVID-19 pandemic: A qualitative study. Nurs Crit Care. 2021 Sep;26(5):397-406. doi: 10.1111/nicc.12589. Epub 2021 Jan 5. PMID 33401340
- [Background] Ferrara M, Funaro MC, Vacca F, Kusmann F, Tedeschini E, Galeazzi GM, Scattoni ML, Starace F. The cost of caring during recent epidemics: a rapid review of risk factors, psychological manifestations, and strategies for its treatment. Ann Ist Super Sanita. 2021 Jan-Mar;57(1):7-17. doi: 10.4415/ANN_21_01_02. PMID 33797399
- [Background] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Background] Fox KC, Dixon ML, Nijeboer S, Girn M, Floman JL, Lifshitz M, Ellamil M, Sedlmeier P, Christoff K. Functional neuroanatomy of meditation: A review and meta-analysis of 78 functional neuroimaging investigations. Neurosci Biobehav Rev. 2016 Jun;65:208-28. doi: 10.1016/j.neubiorev.2016.03.021. Epub 2016 Mar 28. PMID 27032724
- [Background] Friborg O, Hjemdal O, Rosenvinge JH, Martinussen M. A new rating scale for adult resilience: what are the central protective resources behind healthy adjustment? Int J Methods Psychiatr Res. 2003;12(2):65-76. doi: 10.1002/mpr.143. PMID 12830300
- [Background] Gomez-Salgado J, Arias-Ulloa CA, Ortega-Moreno M, Garcia-Iglesias JJ, Escobar-Segovia K, Ruiz-Frutos C. Sense of Coherence in Healthcare Workers During the COVID-19 Pandemic in Ecuador: Association With Work Engagement, Work Environment and Psychological Distress Factors. Int J Public Health. 2022 Dec 5;67:1605428. doi: 10.3389/ijph.2022.1605428. eCollection 2022. PMID 36545403
- [Background] Garcia CL, Abreu LC, Ramos JLS, Castro CFD, Smiderle FRN, Santos JAD, Bezerra IMP. Influence of Burnout on Patient Safety: Systematic Review and Meta-Analysis. Medicina (Kaunas). 2019 Aug 30;55(9):553. doi: 10.3390/medicina55090553. PMID 31480365
- [Background] Goh YS, Ow Yong QYJ, Chen TH, Ho SHC, Chee YIC, Chee TT. The Impact of COVID-19 on nurses working in a University Health System in Singapore: A qualitative descriptive study. Int J Ment Health Nurs. 2021 Jun;30(3):643-652. doi: 10.1111/inm.12826. Epub 2020 Dec 5. PMID 33280242
- [Background] Gonzalez-Gil MT, Gonzalez-Blazquez C, Parro-Moreno AI, Pedraz-Marcos A, Palmar-Santos A, Otero-Garcia L, Navarta-Sanchez MV, Alcolea-Cosin MT, Arguello-Lopez MT, Canalejas-Perez C, Carrillo-Camacho ME, Casillas-Santana ML, Diaz-Martinez ML, Garcia-Gonzalez A, Garcia-Perea E, Martinez-Marcos M, Martinez-Martin ML, Palazuelos-Puerta MDP, Sellan-Soto C, Oter-Quintana C. Nurses' perceptions and demands regarding COVID-19 care delivery in critical care units and hospital emergency services. Intensive Crit Care Nurs. 2021 Feb;62:102966. doi: 10.1016/j.iccn.2020.102966. Epub 2020 Oct 28. PMID 33172732
- [Background] Gordon JM, Magbee T, Yoder LH. The experiences of critical care nurses caring for patients with COVID-19 during the 2020 pandemic: A qualitative study. Appl Nurs Res. 2021 Jun;59:151418. doi: 10.1016/j.apnr.2021.151418. Epub 2021 Mar 11. PMID 33947512
- [Background] Guo YF, Cross W, Plummer V, Lam L, Luo YH, Zhang JP. Exploring resilience in Chinese nurses: a cross-sectional study. J Nurs Manag. 2017 Apr;25(3):223-230. doi: 10.1111/jonm.12457. Epub 2017 Feb 6. PMID 28164403
- [Background] Harper CA, Satchell LP, Fido D, Latzman RD. Functional Fear Predicts Public Health Compliance in the COVID-19 Pandemic. Int J Ment Health Addict. 2021;19(5):1875-1888. doi: 10.1007/s11469-020-00281-5. Epub 2020 Apr 27. PMID 32346359
- [Background] Hart PL, Brannan JD, De Chesnay M. Resilience in nurses: an integrative review. J Nurs Manag. 2014 Sep;22(6):720-34. doi: 10.1111/j.1365-2834.2012.01485.x. Epub 2012 Nov 2. PMID 25208943
- [Background] Hoedl M, Bauer S, Eglseer D. Influence of nursing staff working hours on stress levels during the COVID-19 pandemic: A cross-sectional online survey. HeilberufeScience. 2021;12(3-4):92-98. doi: 10.1007/s16024-021-00354-y. Epub 2021 Sep 10. PMID 34522573
- [Background] Hoge EA, Bui E, Goetter E, Robinaugh DJ, Ojserkis RA, Fresco DM, Simon NM. Change in Decentering Mediates Improvement in Anxiety in Mindfulness-Based Stress Reduction for Generalized Anxiety Disorder. Cognit Ther Res. 2015 Apr;39(2):228-235. doi: 10.1007/s10608-014-9646-4. Epub 2014 Oct 14. PMID 28316355
- [Background] Hummel S, Oetjen N, Du J, Posenato E, Resende de Almeida RM, Losada R, Ribeiro O, Frisardi V, Hopper L, Rashid A, Nasser H, Konig A, Rudofsky G, Weidt S, Zafar A, Gronewold N, Mayer G, Schultz JH. Mental Health Among Medical Professionals During the COVID-19 Pandemic in Eight European Countries: Cross-sectional Survey Study. J Med Internet Res. 2021 Jan 18;23(1):e24983. doi: 10.2196/24983. PMID 33411670
- [Background] Jorgensen F, Bor A, Rasmussen MS, Lindholt MF, Petersen MB. Pandemic fatigue fueled political discontent during the COVID-19 pandemic. Proc Natl Acad Sci U S A. 2022 Nov 29;119(48):e2201266119. doi: 10.1073/pnas.2201266119. Epub 2022 Nov 21. PMID 36413499
- [Background] Karimi Khordeh N, Dehvan F, Dalvand S, Repisti S, Ghanei Gheshlagh R. The COVID-19 fear, anxiety, and resilience among emergency nurses. Front Psychol. 2022 Sep 2;13:999111. doi: 10.3389/fpsyg.2022.999111. eCollection 2022. PMID 36118421
- [Background] Kriakous SA, Elliott KA, Lamers C, Owen R. The Effectiveness of Mindfulness-Based Stress Reduction on the Psychological Functioning of Healthcare Professionals: a Systematic Review. Mindfulness (N Y). 2021;12(1):1-28. doi: 10.1007/s12671-020-01500-9. Epub 2020 Sep 24. PMID 32989406
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Labrague LJ. Pandemic fatigue and clinical nurses' mental health, sleep quality and job contentment during the covid-19 pandemic: The mediating role of resilience. J Nurs Manag. 2021 Oct;29(7):1992-2001. doi: 10.1111/jonm.13383. Epub 2021 Jun 9. PMID 34018270
- [Background] Labrague LJ. Psychological resilience, coping behaviours and social support among health care workers during the COVID-19 pandemic: A systematic review of quantitative studies. J Nurs Manag. 2021 Oct;29(7):1893-1905. doi: 10.1111/jonm.13336. Epub 2021 Apr 28. PMID 33843087
- [Background] Labrague LJ, Ballad CA. Lockdown fatigue among college students during the COVID-19 pandemic: Predictive role of personal resilience, coping behaviors, and health. Perspect Psychiatr Care. 2021 Oct;57(4):1905-1912. doi: 10.1111/ppc.12765. Epub 2021 Mar 17. PMID 33728666
- [Background] Labrague LJ, De Los Santos JAA. Prevalence and predictors of coronaphobia among frontline hospital and public health nurses. Public Health Nurs. 2021 May;38(3):382-389. doi: 10.1111/phn.12841. Epub 2020 Nov 23. PMID 33226158
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Leng M, Wei L, Shi X, Cao G, Wei Y, Xu H, Zhang X, Zhang W, Xing S, Wei H. Mental distress and influencing factors in nurses caring for patients with COVID-19. Nurs Crit Care. 2021 Mar;26(2):94-101. doi: 10.1111/nicc.12528. Epub 2020 Jul 27. PMID 33448567
- [Background] Liu Q, Luo D, Haase JE, Guo Q, Wang XQ, Liu S, Xia L, Liu Z, Yang J, Yang BX. The experiences of health-care providers during the COVID-19 crisis in China: a qualitative study. Lancet Glob Health. 2020 Jun;8(6):e790-e798. doi: 10.1016/S2214-109X(20)30204-7. Epub 2020 Apr 29. PMID 32573443
- [Background] Lin L, He G, Yan J, Gu C, Xie J. The Effects of a Modified Mindfulness-Based Stress Reduction Program for Nurses: A Randomized Controlled Trial. Workplace Health Saf. 2019 Mar;67(3):111-122. doi: 10.1177/2165079918801633. Epub 2018 Oct 29. PMID 30370837
- [Background] Liu Y, Xian JS, Wang R, Ma K, Li F, Wang FL, Yang X, Mu N, Xu K, Quan YL, Wang S, Lai Y, Yang CY, Li T, Zhang Y, Tan B, Feng H, Chen TN, Wang LH. Factoring and correlation in sleep, fatigue and mental workload of clinical first-line nurses in the post-pandemic era of COVID-19: A multi-center cross-sectional study. Front Psychiatry. 2022 Aug 25;13:963419. doi: 10.3389/fpsyt.2022.963419. eCollection 2022. PMID 36090368
- [Background] Lazaro-Perez C, Martinez-Lopez JA, Gomez-Galan J, Lopez-Meneses E. Anxiety About the Risk of Death of Their Patients in Health Professionals in Spain: Analysis at the Peak of the COVID-19 Pandemic. Int J Environ Res Public Health. 2020 Aug 15;17(16):5938. doi: 10.3390/ijerph17165938. PMID 32824258
- [Background] Luthar SS, Cicchetti D, Becker B. The construct of resilience: a critical evaluation and guidelines for future work. Child Dev. 2000 May-Jun;71(3):543-62. doi: 10.1111/1467-8624.00164. PMID 10953923
- [Background] Lutz A, Jha AP, Dunne JD, Saron CD. Investigating the phenomenological matrix of mindfulness-related practices from a neurocognitive perspective. Am Psychol. 2015 Oct;70(7):632-58. doi: 10.1037/a0039585. PMID 26436313
- [Background] Majumdar P, Biswas A, Sahu S. COVID-19 pandemic and lockdown: cause of sleep disruption, depression, somatic pain, and increased screen exposure of office workers and students of India. Chronobiol Int. 2020 Aug;37(8):1191-1200. doi: 10.1080/07420528.2020.1786107. Epub 2020 Jul 13. PMID 32660352
- [Background] Marotta M, Gorini F, Parlanti A, Berti S, Vassalle C. Effect of Mindfulness-Based Stress Reduction on the Well-Being, Burnout and Stress of Italian Healthcare Professionals during the COVID-19 Pandemic. J Clin Med. 2022 May 31;11(11):3136. doi: 10.3390/jcm11113136. PMID 35683520
- [Background] Mealer M, Jones J, Moss M. A qualitative study of resilience and posttraumatic stress disorder in United States ICU nurses. Intensive Care Med. 2012 Sep;38(9):1445-51. doi: 10.1007/s00134-012-2600-6. Epub 2012 May 23. PMID 22618093
- [Background] Mealer M, Jones J, Newman J, McFann KK, Rothbaum B, Moss M. The presence of resilience is associated with a healthier psychological profile in intensive care unit (ICU) nurses: results of a national survey. Int J Nurs Stud. 2012 Mar;49(3):292-9. doi: 10.1016/j.ijnurstu.2011.09.015. Epub 2011 Oct 5. PMID 21974793
- [Background] Mealer M, Conrad D, Evans J, Jooste K, Solyntjes J, Rothbaum B, Moss M. Feasibility and acceptability of a resilience training program for intensive care unit nurses. Am J Crit Care. 2014 Nov;23(6):e97-105. doi: 10.4037/ajcc2014747. PMID 25362680
- [Background] Mehta DH, Perez GK, Traeger L, Park ER, Goldman RE, Haime V, Chittenden EH, Denninger JW, Jackson VA. Building Resiliency in a Palliative Care Team: A Pilot Study. J Pain Symptom Manage. 2016 Mar;51(3):604-8. doi: 10.1016/j.jpainsymman.2015.10.013. Epub 2015 Nov 6. PMID 26550936
- [Background] Melnyk BM, Kelly SA, Stephens J, Dhakal K, McGovern C, Tucker S, Hoying J, McRae K, Ault S, Spurlock E, Bird SB. Interventions to Improve Mental Health, Well-Being, Physical Health, and Lifestyle Behaviors in Physicians and Nurses: A Systematic Review. Am J Health Promot. 2020 Nov;34(8):929-941. doi: 10.1177/0890117120920451. Epub 2020 Apr 27. PMID 32338522
- [Background] Murphy JFA. Pandemic Fatigue. Ir Med J. 2020 Jun 11;113(6):90. No abstract available. PMID 32816425
- [Background] Nasirizad Moghadam K, Chehrzad MM, Reza Masouleh S, Maleki M, Mardani A, Atharyan S, Harding C. Nursing physical workload and mental workload in intensive care units: Are they related? Nurs Open. 2021 Jul;8(4):1625-1633. doi: 10.1002/nop2.785. Epub 2021 Feb 17. PMID 33596333
- [Background] Othman SY, Hassan NI, Mohamed AM. Effectiveness of mindfulness-based interventions on burnout and self-compassion among critical care nurses caring for patients with COVID-19: a quasi-experimental study. BMC Nurs. 2023 Sep 6;22(1):305. doi: 10.1186/s12912-023-01466-8. PMID 37674145
- [Background] Perez V, Menendez-Crispin EJ, Sarabia-Cobo C, de Lorena P, Fernandez-Rodriguez A, Gonzalez-Vaca J. Mindfulness-Based Intervention for the Reduction of Compassion Fatigue and Burnout in Nurse Caregivers of Institutionalized Older Persons with Dementia: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Sep 11;19(18):11441. doi: 10.3390/ijerph191811441. PMID 36141714
- [Background] Placzek M, Friede T. Clinical trials with nested subgroups: Analysis, sample size determination and internal pilot studies. Stat Methods Med Res. 2018 Nov;27(11):3286-3303. doi: 10.1177/0962280217696116. Epub 2017 Mar 14. PMID 29298604
- [Background] Reger MA, Piccirillo ML, Buchman-Schmitt JM. COVID-19, Mental Health, and Suicide Risk Among Health Care Workers: Looking Beyond the Crisis. J Clin Psychiatry. 2020 Aug 4;81(5):20com13381. doi: 10.4088/JCP.20com13381. No abstract available. PMID 32757506
- [Background] Ren HF, Chen FJ, He LX, Liu CQ, Liu YY, Huang YJ, Han H, Fu S, Zhang MG, Jiang Y. Nursing allocation in isolation wards of COVID-19 designated hospitals: a nationwide study in China. BMC Nurs. 2022 Jan 19;21(1):23. doi: 10.1186/s12912-021-00795-w. PMID 35042486
- [Background] Resnick B. Covid-19 lessons learned from the voices of our geriatric nurses: Leadership, resilience, and heroism. Geriatr Nurs. 2020 Jul-Aug;41(4):357-359. doi: 10.1016/j.gerinurse.2020.06.008. Epub 2020 Jun 18. No abstract available. PMID 32680676
- [Background] Sallon S, Katz-Eisner D, Yaffe H, Bdolah-Abram T. Caring for the Caregivers: Results of an Extended, Five-component Stress-reduction Intervention for Hospital Staff. Behav Med. 2017 Jan-Mar;43(1):47-60. doi: 10.1080/08964289.2015.1053426. Epub 2015 Nov 7. PMID 26548543
- [Background] Salzberger B, Buder F, Lampl B, Ehrenstein B, Hitzenbichler F, Holzmann T, Schmidt B, Hanses F. Epidemiology of SARS-CoV-2. Infection. 2021 Apr;49(2):233-239. doi: 10.1007/s15010-020-01531-3. Epub 2020 Oct 8. PMID 33034020
- [Background] Schroeder DA, Stephens E, Colgan D, Hunsinger M, Rubin D, Christopher MS. A Brief Mindfulness-Based Intervention for Primary Care Physicians: A Pilot Randomized Controlled Trial. Am J Lifestyle Med. 2016 Feb 4;12(1):83-91. doi: 10.1177/1559827616629121. eCollection 2018 Jan-Feb. PMID 30202383
- [Background] Senders A, Hanes D, Bourdette D, Carson K, Marshall LM, Shinto L. Impact of mindfulness-based stress reduction for people with multiple sclerosis at 8 weeks and 12 months: A randomized clinical trial. Mult Scler. 2019 Jul;25(8):1178-1188. doi: 10.1177/1352458518786650. Epub 2018 Jul 9. PMID 29985095
- [Background] Serrano-Ripoll MJ, Meneses-Echavez JF, Ricci-Cabello I, Fraile-Navarro D, Fiol-deRoque MA, Pastor-Moreno G, Castro A, Ruiz-Perez I, Zamanillo Campos R, Goncalves-Bradley DC. Impact of viral epidemic outbreaks on mental health of healthcare workers: a rapid systematic review and meta-analysis. J Affect Disord. 2020 Dec 1;277:347-357. doi: 10.1016/j.jad.2020.08.034. Epub 2020 Aug 23. PMID 32861835
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Sun N, Wei L, Shi S, Jiao D, Song R, Ma L, Wang H, Wang C, Wang Z, You Y, Liu S, Wang H. A qualitative study on the psychological experience of caregivers of COVID-19 patients. Am J Infect Control. 2020 Jun;48(6):592-598. doi: 10.1016/j.ajic.2020.03.018. Epub 2020 Apr 8. PMID 32334904
- [Background] Tang X, Pei Y, Wang X, Jiang L, Liu P, Chen Y, Meng Z. Mental health and fatigue status of the medical workforce during the COVID-19 outbreak in the Yangzhou city, China. Front Psychiatry. 2022 Oct 17;13:1018069. doi: 10.3389/fpsyt.2022.1018069. eCollection 2022. PMID 36325526
- [Background] Tang YY, Holzel BK, Posner MI. The neuroscience of mindfulness meditation. Nat Rev Neurosci. 2015 Apr;16(4):213-25. doi: 10.1038/nrn3916. Epub 2015 Mar 18. PMID 25783612
- [Background] Umbetkulova S, Kanderzhanova A, Foster F, Stolyarova V, Cobb-Zygadlo D. Mental Health Changes in Healthcare Workers During COVID-19 Pandemic: A Systematic Review of Longitudinal Studies. Eval Health Prof. 2024 Mar;47(1):11-20. doi: 10.1177/01632787231165076. Epub 2023 May 4. PMID 37143216
- [Background] Usher K, Jackson D, Durkin J, Gyamfi N, Bhullar N. Pandemic-related behaviours and psychological outcomes; A rapid literature review to explain COVID-19 behaviours. Int J Ment Health Nurs. 2020 Dec;29(6):1018-1034. doi: 10.1111/inm.12790. Epub 2020 Oct 13. PMID 32860475
- [Background] Wang Y, Tang L, Li L. Work engagement and associated factors among healthcare professionals in the post-pandemic era: a cross-sectional study. Front Public Health. 2023 Jul 27;11:1173117. doi: 10.3389/fpubh.2023.1173117. eCollection 2023. PMID 37575106
- [Background] Wax RS, Christian MD. Practical recommendations for critical care and anesthesiology teams caring for novel coronavirus (2019-nCoV) patients. Can J Anaesth. 2020 May;67(5):568-576. doi: 10.1007/s12630-020-01591-x. Epub 2020 Feb 12. PMID 32052373
- [Background] White L. Mindfulness in nursing: an evolutionary concept analysis. J Adv Nurs. 2014 Feb;70(2):282-94. doi: 10.1111/jan.12182. Epub 2013 Jun 16. PMID 23772683
- [Background] Wielgosz J, Goldberg SB, Kral TRA, Dunne JD, Davidson RJ. Mindfulness Meditation and Psychopathology. Annu Rev Clin Psychol. 2019 May 7;15:285-316. doi: 10.1146/annurev-clinpsy-021815-093423. Epub 2018 Dec 10. PMID 30525995
- [Background] Windle G, Bennett KM, Noyes J. A methodological review of resilience measurement scales. Health Qual Life Outcomes. 2011 Feb 4;9:8. doi: 10.1186/1477-7525-9-8. PMID 21294858
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Zhan YX, Zhao SY, Yuan J, Liu H, Liu YF, Gui LL, Zheng H, Zhou YM, Qiu LH, Chen JH, Yu JH, Li SY. Prevalence and Influencing Factors on Fatigue of First-line Nurses Combating with COVID-19 in China: A Descriptive Cross-Sectional Study. Curr Med Sci. 2020 Aug;40(4):625-635. doi: 10.1007/s11596-020-2226-9. Epub 2020 Aug 29. PMID 32767264
- [Derived] Hsieh CW, Sun WN, Chiang HY, Weng SF, Hsu YF, Yu E, Hsu HT. Effectiveness of an online mindfulness-based stress reduction program for nurses in high-stress occupational settings during the COVID-19 pandemic. Appl Nurs Res. 2026 Feb;87:152032. doi: 10.1016/j.apnr.2025.152032. Epub 2025 Nov 27. PMID 41578985